CLINICAL TRIAL: NCT07080242
Title: A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BL-M14D1 in Subjects With Locally Advanced or Metastatic Small Cell Lung Cancer and Other Neuroendocrine Neoplasms
Brief Title: Evaluating BL-M14D1 in Subjects With Locally Advanced or Metastatic Small Cell Lung Cancer and Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-M14D1-ST-101
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer Metastatic or Locally Advanced; Neuroendocrine Cancer; Metastatic or Locally Advanced Neuroendocrine Prostate Cancer; Metastatic or Locally Advanced Poorly Differentiated Gastroenteropancreatic Neuroendocrine Carcinoma; Metastatic or Locally Advanced Merkel Cell Carcinoma; Locally Advanced or Metastatic Large Cell Neuroendocrine Carcinoma of the Lung; Metastatic or Locally Advanced Extrapulmonary Neuroendocrine Carcinoma; Poorly Differentiated and/or High Grade Neuroendocrine Neoplasms With Evidence of DLL3 Expression
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental BL-M14D1 administered Day 1 per cycle (Experimental): BL-M14D1 will be administered on Day 1 by intravenous (IV) infusion every 3 weeks
  Interventions: Drug: BL-M14D1

INTERVENTIONS:
Drug: BL-M14D1 — BL-M14D1 will be administered on D1 every 3 weeks.

SUMMARY:
The objective of this study is to evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BL-M14D1 in Subjects with locally Advanced or Metastatic Small Cell Lung Cancer and Other Neuroendocrine Neoplasms

DETAILED DESCRIPTION:
A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BL-M14D1 in Subjects With Locally Advanced or Metastatic Small Cell Lung Cancer and Other Neuroendocrine Neoplasms

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form voluntarily and agreed to follow the trial requirements
2. Age ≥18 years
3. Participant weighs more than 40 kg
4. Life expectancy of ≥3 months
5. Documented locally advanced or metastatic SCLC, large cell neuroendocrine cancer of the lung (LCNEC), neuroendocrine prostate cancer (NEPC), poorly differentiated gastroenteropancreatic neuroendocrine carcinomas (GEP-NEC) or other extrapulmonary neuroendocrine carcinomas (EP-NECs), Merkel cell carcinoma (MCC), or other poorly differentiated and/or high-grade neuroendocrine neoplasms with evidence of DLL3 expression who have failed at least 1 line of standard therapy in the advanced/metastatic setting or are unable to receive standard treatment Notes: For SCLC, the participant must have failed at least 1 line of platinum therapy in the advanced/metastatic setting. No prior topoisomerase inhibitor-based ADC therapy is permitted. In the dose expansion part, Cohort 6 (DLL3-Positive NEN Subgroup): participants will be eligible based on documented positive DLL3 expression.
6. Agree to provide archival tumor samples (formalin-fixed paraffin-embedded [FFPE] tissue block or 6-12 slides of 5-μm thickness) from primary or metastatic sites:

   1. In dose escalation and dose finding: archival tissue should be obtained within 2 years or FFPE block from fresh biopsy. If no archival tissue is available, a fresh tissue biopsy is required
   2. In dose expansion: an FFPE block from fresh biopsy or archival tissue (within 6 months) is required NOTE: If no archival tissue is available and, a fresh tissue biopsy is clinically contraindicated, please consult the sponsor.
7. At least one measurable lesion based on RECIST (Response Evaluation Criteria in Solid Tumors) v1.1
8. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1
9. Toxicity of previous antitumor therapy has returned to Grade ≤1 as defined by National Cancer Institute (NCI) CTCAE v5.0, except for alopecia and endocrinopathies controlled by replacement therapy
10. No serious cardiac dysfunction and left ventricular ejection fraction ≥50%
11. Adequate organ function, defined as:

    1. Marrow function: Absolute neutrophil count (ANC) ≥1.5×10^9/, platelet count

       ≥100×10^9/L, hemoglobin (Hb) ≥9.0 g/dL (blood transfusion, platelet transfusion, erythropoietin (EPO), hematopoiesis agents (such as thrombopoietin [TPO]), and granulocyte colony-stimulating factor [G-CSF] use are not allowed 1 week prior to screening)
    2. Hepatic function: Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) (≤3×ULN for participants with liver metastasis at baseline), AST and alanine aminotransferase (ALT) without liver metastasis ≤3.0×ULN, AST and ALT with liver metastasis ≤5.0×ULN NOTE: For participants with Gilbert's syndrome, TBIL ≤3.0×ULN in the absence of liver metastases.
    3. Renal function: Creatinine (Cr) clearance ≥60 mL/minute (Cockcroft-Gault equation) or estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2 (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation)
12. Coagulation parameters: International normalized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (aPTT) ≤1.5×ULN, unless receiving anticoagulation therapy with PT and aPTT levels within the intended therapeutic range
13. Urine protein ≤2+ or ≤1000 mg/24 hours
14. Sexually active fertile participants and their partners must agree to use highly effective methods of contraception (defined in Appendix D) during the course of the study and after the last dose of study treatment (7 months for women of childbearing potential [WOCP] and 4 months for men). An additional contraceptive method, such as a barrier method (eg, condom), is recommended.
15. WOCBP must have a negative serum pregnancy test at screening and must be nonlactating. Female participants are considered WOCBP unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman >45 years old in the absence of other biological or physiological causes). In addition, females <55 years old must have a serum follicle stimulating hormone (FSH) level >40 mIU/mL to confirm menopause.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, , targeted therapy (including small molecule inhibitor of tyrosine kinase), and other antitumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; radical radiotherapy, major surgery within 4 weeks prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration; oral fluorouracil drugs such as tegafur, capecitabine, or palliative radiotherapy within 2 weeks prior to initial administration.
2. Participants who have received prior topoisomerase inhibitor-based ADC therapy
3. Concomitant use of strong inhibitors and inducers of any CYP enzyme or transporter system within 2 weeks prior to the first administration and throughout all parts of the study
4. Participants with history of severe heart disease, such as symptomatic (CHF) ≥Grade 2 (CTCAE v5.0), New York Heart Association (NYHA) ≥Grade 2 heart failure at any time, history of myocardial infarction or unstable angina pectoris within 6 months before enrollment
5. Participants with prolonged QT interval corrected (Fridericia formula (QTcF >470 msec), complete left bundle branch block, Grade 3 atrioventricular block, or a history of additional risk factors for Torsades de Pointes (TdP); eg, heart failure as defined in Exclusion Criterion 4, chronic or recurrent hypokalemia that requires medical intervention, congenital long QT syndrome, family history of long QT syndrome) or any current concomitant medication known to prolong the QT/QTc interval or cause TdP.
6. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease, and Hashimoto's thyroiditis, etc. Participants with skin diseases that do not require systemic treatment (such as vitiligo, psoriasis), well-controlled type 1 diabetes, or hypothyroidism are permitted. For autoimmune conditions that are active but stable and low grade on systemic therapy, discussion with the medical monitor is required prior to screening.
7. Participants with other prior or concurrent malignancies except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after adequate resection, or other malignancy treated with curative intent with a disease-free interval of at least 3 years
8. Participants with poorly controlled hypertension by 2 types of antihypertensive drugs (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg)
9. Participants with advanced/ clinically significant lung diseases, such as poorly controlled chronic obstructive pulmonary disease (COPD) and asthma, restrictive lung disease, pulmonary hypertension etc.
10. Participants who have a history of noninfectious ILD/pneumonitis that required treatment with steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
11. Participants with stroke or transient ischemic attack (TIA) within 6 months before screening
12. Participants with a thromboembolic event (eg, deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 6 months before screening except for those who are clinically stable and receiving treatment with adequate anticoagulant therapy for at least 3 weeks before screening
13. Participants with primary neoplasms in the (CNS), active or untreated CNS metastases or carcinomatous meningitis should be excluded. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks and have no radiological evidence of new or enlarging brain metastases and no requirements for corticosteroids 14 days prior to screening.
14. Participants with preexisting Grade ≥2 peripheral neuropathy
15. Participants who have a history of anaphylaxis or severe hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of BL-M14D1
16. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation
17. Participants who are receiving treatment with systemic glucocorticoids >10 mg/day equivalent of prednisone, except for the treatment of COPD, antiemetic, infusion reactions; however, treatment with low dose glucocorticoids (≤10 mg/day equivalent of prednisone) is permitted. The use of topical, inhaled, and locally injected steroids is permitted
18. Participants with known human immunodeficiency virus infection (HIV Ab positive). Subjects are allowed to participate if all of the following criteria are met: (1) Undetectable HIV RNA and CD4 count ≥350 cells/μL at Screening, (2) No AIDS-defining opportunistic infection within 12 months prior to screening, (3) On stable antiretroviral therapy (ART) for at least 4 weeks prior to Screening with projected continuation of ART as clinically indicated while on the study
19. Participants with active hepatitis B virus (HBV) infection (positive HBsAg test). Participants with chronic inactive HBV infection are eligible if they meet all of the following criteria:

    1. Have a HBV DNA viral load ≤ 500 IU/mL
    2. Normal AST and ALT, OR if liver metastasis is present, has AST and ALT < 3 × ULN which are not attributed to HIV infection
    3. Are on antiviral treatment, as clinically indicated.
20. Participants with active hepatitis C virus (HCV) infection (HCV antibody positive and HCV RNA > the lower limit of detection). Participants with a positive anti-HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
21. Participants with active or latent tuberculosis
22. Participants with active infections requiring IV antibiotic, antiviral, or antifungal treatment, such as severe pneumonia, bacteremia, sepsis, etc., within 1 week prior to first dose of study treatment. Subjects on stable oral antimicrobials with no clinical or laboratory evidence of active infection are eligible.
23. Participated in another clinical trial within 4 weeks prior to first dose of study treatment
24. Participants who are pregnant or breastfeeding, or planning to become pregnant during the study
25. Other conditions that the Investigator or Sponsor believes are not suitable for participating in this clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants with Dose-limiting toxicities | 1 Year
  A DLT is defined as any of the following events:
  Toxicity that results in a >14-day delay in treatment
  * Hematologic toxicities:
    * Grade 4 neutrophil count decreased lasting >7 days
    * Grade ≥3 febrile neutropenia of any duration
    * Grade ≥3 platelet count decreased with clinically significant hemorrhage
  * Nonhematologic toxicities:
    * Death not related to disease progression or extraneous cause
    * Hy's law cases
    * Grade ≥3 nonhematologic toxicities, except for:
      * Grade 3 nausea/vomiting or diarrhea for less than 72 hours with adequate antiemetic and other supportive care
      * Grade 3 fatigue for less than 1 week
      * Grade ≥3 electrolyte abnormality that lasts up to 72 hours, is not clinically complicated, and resolves spontaneously or responds to conventional medical interventions
      * Grade ≥3 amylase or lipase that is not associated with symptoms or clinical manifestations of pancreatitis
Participants with Serious Adverse Events (SAEs) and treatment-emergent adverse events (TEAEs) | 1 Year
  Measuring the number of patients with serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs)
Participants with abnormal physical examination findings | 1 Year
  Measure the number of participants with abnormal physical examination findings.
Participants with ability to care for themselves, daily activity, and physical activity | 1 Year
  Measure the change in participants with Eastern Clinical Oncology Group (ECOG) Scale of Performance Status. The scale is 0-4 with 0 being the fully active (best outcome) and 4 being completely disabled (worst outcome)
Participants with abnormal ECG and ECHO/MUGA reading | 1 Year
  Patients with abnormal ECG parameters (including the change from-baseline ECG parameters: heart rate [HR]; PR; QTcF; and QRS intervals [∆HR, ∆PR, ∆QTcF, and ∆QRS]), and ECHO/MUGA findings
Participants with abnormal lab results | 1 Year
  Measure the number of participants with abnormal clinical laboratory values
To determine the maximum tolerated dose (MTD) if reached or maximum administered dose (MAD) and two or more recommended doses for expansion (RDEs) of BL-M05D1 in metastatic or unresectable tumors | 1 Year
  The actual number of subjects enrolled and dose levels to be explored in this study will depend on the MTD and/or RDE based on DLTs reported during the DLT observation period.

SECONDARY OUTCOMES:
Cmax of BL-M14D1 | 1 Year
  Calculate maximum (peak) observed concentration of BL-M14D1
Cmax of anti-DLL3 antibodies | 1 Year
  Calculate maximum (peak) observed concentration of anti-BL-DLL3 antibodies
Cmax of free payload ED-04 | 1 Year
  Calculate maximum (peak) observed concentration of free payload ED-04
Tmax of BL-M14D1 | 1 Year
  Calculate time of maximum observed concentration of BL-M14D1
Tmax of anti-DLL3 antibodies | 1 Year
  Calculate time of maximum observed concentration of anti-DLL3 antibodies
Tmax of free payload ED-04 | 1 Year
  Calculate time of maximum observed concentration of free payload ED-04
AUC(0-8) of BL-M05D1 | 1 Year
  Calculate area under the serum concentration-time curve of BL-M05D1 from time 0 to 8 hours
AUC(0-8) of anti-DLL3 antibodies | 1 Year
  Calculate area under the serum concentration-time curve of anti-DLL3 antibodies from time 0 to 8 hours
AUC(0-8) of free payload ED-04 | 1 Year
  Calculate area under the serum concentration-time curve of free payload ED-04 from time 0 to 8 hours
AUC(last) of BL-M14D1 | 1 Year
  Calculate area under the serum concentration-time curve up of BL-M05D1 to the last quantifiable time 0 to 8 hours
AUC(last) of anti-DLL3 antibodies | 1 Year
  Calculate area under the serum concentration-time curve up of anti-BL-M05D1 antibodies to the last quantifiable time 0 to 8 hours
AUC(last) of free payload ED-04 | 1 Year
  Calculate area under the serum concentration-time curve up of free payload ED-04 to the last quantifiable time
Overall Response Rate (ORR) | 1 Year
  To assess the clinical efficacy of BL-M14D1 as measured by ORR using RECIST criteria v 1.1
Disease Control Rate (DCR) | 1 Year
  To assess the clinical efficacy of BL-M14D1 as measured by DCR using RECIST criteria v 1.1
Time To Response (TTR) | 1 Year
  To assess the clinical efficacy of BL-M05D1 as measured by TTR using RECIST criteria v 1.1
Progression-Free Survival (PFS) | 1 Year
  To assess the clinical efficacy of BL-M14D1 as measured by PFS using RECIST criteria v 1.1
Overall Survival (OS) | 1 Year
  To assess the clinical efficacy of BL-M14D1 as measured by OS using RECIST criteria v 1.1
Duration of response (DoR) | 1 Year
  To assess the clinical efficacy of BL-M14D1 as measured by DoR using RECIST criteria v 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Jain, Study Director — SystImmune Inc.
Locations (20):
- United States (20):
  - Valkyrie Clinical Trials, Los Angeles, California
  - UCLA, Los Angeles, California
  - UCSF- San Francisco (Helen Diller Family Comprehensive Cancer Center), San Francisco, California
  - University of Colorado - Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Emory Winship, Atlanta, Georgia
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - John Theurer Cancer Center-Hackensack, Hackensack, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University, Columbus, Ohio
  - Providence Cancer Institute, Portland, Oregon
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - NEXT Dallas, Dallas, Texas
  - START Dallas- Fort Worth, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Houston, Houston, Texas
  - START- San Antonio, San Antonio, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
  - University of Washington/Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No